CLINICAL TRIAL: NCT05197374
Title: Studying The Effect of Estradiol Pretreatment on Follicular Synchronization and Intracytoplasmic Sperm Injection (ICSI) Outcome in Antagonist Cycles
Brief Title: Effect of Estradiol Pretreatment on Antagonist ICSI Cycles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0106351
Record Dates: First submitted 2022-01-05; First posted 2022-01-19 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female | interventions — Estradiol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Cases who received estradiol pretreatment then underwent ICSI.
  Interventions: Drug: Estradiol Valerate 4mg
- group 2 (No Intervention): Cases who underwent ICSI directly without receiving any pretreatment

INTERVENTIONS:
Drug: Estradiol Valerate 4mg — Estradiol valerate 2 mg (two tablet once daily) started 5 days before expected menses (or 7 days after ovulation of previous cycle). After start of menses, estradiol pretreatment was stopped and controlled ovarian stimulation started.
  Other Names: Progynova
  Arms: Group 1

SUMMARY:
Depended on the hypothesis that growth asynchrony of antral follicles is a consequence of the gradual follicle stimulating hormone (FSH) elevation that occurs during the late luteal phase, the aim of this work is to study the effect of estradiol pretreatment on follicular synchronization and intracytoplasmic sperm injection (ICSI) outcome in antagonist cycles

DETAILED DESCRIPTION:
Gonadotropin-releasing hormone antagonist (GnRH-ant) cycles are characterized by higher patient acceptability with more attention being directed to the potential effect of steroid pretreatment to program antagonist protocol cycles, as marked size discrepancies of growing follicles reflect incoordinated maturation of follicular-oocyte complexes and complicates clinical criteria for human chorionic gonadotropin (hCG) administration. This phenomenon is associated with fewer mature oocytes and resulting embryos, which limits sufficient embryo selection for embryo transfer. Indeed, the large number of available embryos represented an important prognostic factor of invitro-fertilization (IVF) outcome, particularly in poor prognosis patients, possibly by increasing the probability that at least one good-quality embryo will be selected for embryo transfer. During COH, a better understanding of follicular development has resulted in the improvement of strategies for ovarian stimulation. This approach represents a potential and more physiological alternative to GnRH agonist or oral contraceptive pills pre-treatment in a trial to synchronize multi-follicular development and improve controlled ovarian hyperstimulation (COH) results. The present study is a randomized controlled trial that investigated whether E2 pre-treatment during the luteal phase affects developmental characteristics of growing follicles during COH. It depended on the hypothesis that growth asynchrony of antral follicles is a consequence of the gradual FSH elevation that occurs during the late luteal phase, thus testing for detection of the effect of luteal estradiol on follicular synchronization and its effect on ICSI outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Women age 20-37 years.
2. Anti-mullerian (AMH) level greater than 1.2 ng/ml.
3. Body mass index between 18 and 29 kg/m2.
4. Undergoing a first or second ICSI cycles.

Exclusion Criteria:

1. Endometriosis.
2. Uterine disorders such as fibroids and uterine anomalies.
3. Antral follicular counts (AFC) less than 10.
4. Azoospermic males.

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Days of stimulation. | 7-16 days after start of controlled ovarian stimulation.
  number of days from the start of controlled ovarian stimulation on day 2 of menses until the day of hCG administration until day of hCG administration
Total number of gonadotropin ampoules used. | 7-16 days after start of controlled ovarian stimulation.
  number of gonadotropin ampules used from the start of controlled ovarian stimulation on day 2 of menses until the day of hCG administration
Total number of follicles by U/S on day of hCG. | 7-16 days after start of controlled ovarian stimulation.
  number of follicles by ultrasound scan on day of hCG administration
Serum estradiol and progesterone level on day of hCG . | 7-16 days after start of controlled ovarian stimulation.
  serum level of estradiol pg/dl and progesterone ng/dl on day of hCG administration
Endometrial thickness on day of hCG. | 7-16 days after start of controlled ovarian stimulation.
  thickness of endometrium in mm on day of hCG
Number of mature oocytes | 36 hours after oocyte retrieval.
  number of metaphase II oocytes after denudation
Number of good quality embryos. | 3 days after oocyte retrieval.
  number of grade 1 and grade 2 day 3 embryos

SECONDARY OUTCOMES:
Pregnancy rate | 14 days after embryo transfer
  the number of positive pregnancies (defined as serum B-hCG more than 5 miu/ml measured 14 days after embryo transfer) divided by the number of embryo transfer procedures.
Clinical pregnancy rate | 2 weeks after positive pregnancy test
  The number of clinical pregnancies (defined as the presence of a gestational sac with positive heart beat detected by transvaginal ultrasound scan 2 weeks after positive pregnancy test) divided by the number of embryo transfer procedures

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Hebisha, phD, Principal Investigator — Alexandria University
Locations (1):
- IVF center, Alexandria, Egypt

REFERENCES:
- [Background] Devreker F, Pogonici E, De Maertelaer V, Revelard P, Van den Bergh M, Englert Y. Selection of good embryos for transfer depends on embryo cohort size: implications for the 'mild ovarian stimulation' debate. Hum Reprod. 1999 Dec;14(12):3002-8. doi: 10.1093/humrep/14.12.3002. PMID 10601087
- [Background] Opsahl MS, Blauer KL, Black SH, Lincoln SR, Thorsell L, Sherins RJ. The number of embryos available for transfer predicts successful pregnancy outcome in women over 39 years with normal ovarian hormonal reserve testing. J Assist Reprod Genet. 2001 Oct;18(10):551-6. doi: 10.1023/a:1011906024170. PMID 11699127
- [Background] Lee H, Choi HJ, Yang KM, Kim MJ, Cha SH, Yi HJ. Efficacy of luteal estrogen administration and an early follicular Gonadotropin-releasing hormone antagonist priming protocol in poor responders undergoing in vitro fertilization. Obstet Gynecol Sci. 2018 Jan;61(1):102-110. doi: 10.5468/ogs.2018.61.1.102. Epub 2017 Dec 19. PMID 29372156
- [Background] Cedrin-Durnerin I, Guivarc'h-Leveque A, Hugues JN; Groupe d'Etude en Medecine et Endocrinologie de la Reproduction. Pretreatment with estrogen does not affect IVF-ICSI cycle outcome compared with no pretreatment in GnRH antagonist protocol: a prospective randomized trial. Fertil Steril. 2012 Jun;97(6):1359-64.e1. doi: 10.1016/j.fertnstert.2012.02.028. Epub 2012 Mar 28. PMID 22464760
- [Background] Sefrioui O, Madkour A, Kaarouch I, Louanjli N. Luteal estradiol pretreatment of poor and normal responders during GnRH antagonist protocol. Gynecol Endocrinol. 2019 Dec;35(12):1067-1071. doi: 10.1080/09513590.2019.1622086. Epub 2019 May 29. PMID 31142165